CLINICAL TRIAL: NCT06951685
Title: Prospective, Non-randomized, Early Feasibility Clinical Study to Assess the Feasibility of the Novel Xeltis Peripheral Artery Disease (XPAD) Bypass Conduit
Brief Title: Xeltis Peripheral Artery Disease (XPAD) Bypass Conduit Early Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xeltis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEL-CR-15
Record Dates: First submitted 2025-04-11; First posted 2025-04-30 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Artery Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XPAD Bypass Conduit (Experimental)
  Interventions: Device: Xeltis Peripheral Artery Disease (XPAD) Bypass Conduit

INTERVENTIONS:
Device: Xeltis Peripheral Artery Disease (XPAD) Bypass Conduit — The XPAD bypass conduit is a sterile, restorative biodegradable polymer-based vascular graft, consisting of a tubular structure with a 33cm length and 6mm inner diameter. It is comprised of a highly porous polymer matrix and an embedded electropolished nitinol reinforcement layer (Strain Relief System). The XPAD conduit is in a straight configuration and may be implanted above the knee for elective femoral popliteal bypass surgery.

SUMMARY:
A prospective, single arm, non-randomized early feasibility study to evaluate the preliminary safety and performance of the XPAD conduit in patients with peripheral arterial occlusive disease (PAOD), scheduled to undergo elective above-knee femoral popliteal bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with femoral artery occlusion who require elective above-knee femoral popliteal bypass surgery
2. Patient has Rutherford grade 3, 4, or 5 occlusive vascular disease and TASC C or D lesions. Rutherford grade 5 may be included with a wound, ischemia and foot infection (WiFi) classification of up to grade 2, provided there are two outflow vessels with at least one reaching the pedal arch
3. At least 18 years of age at screening
4. Suitable anatomy (assessed by a pre-procedural contrasted CT scan or previous angiogram assessed up to 90 days prior to baseline)
5. Patient has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent
6. Patient has been informed and agrees to pre- and post-procedure follow-up, including follow-up angiography
7. Life expectancy of at least 24 months

Exclusion Criteria:

1. Subject requires, or is scheduled for, a cardiac surgical procedure or a different vascular surgical procedure within 30 days of study procedure.
2. Presence or history of bypass in the diseased limb
3. Subject requires sequential extremity revascularizations or other procedures that require use of additional vascular grafts
4. Stroke or myocardial infarction event within 6 weeks of the procedure or evidence of prior massive stroke (Modified Rankin Scale 3 or above)
5. History of acute arterial occlusion requiring an emergent intervention
6. Severe chronic renal insufficiency (serum creatinine >2.5 mg/dL) or undergoing hemodialysis
7. Previous renal transplant
8. Uncontrolled arterial hypertension (BP >200 mmHg) at 2 successive readings
9. Uncontrolled or poorly controlled diabetes
10. Abnormal blood values that could influence patient recovery and or/ graft hemostasis
11. Reduced liver function, defined as: >2x the upper limit of normal for serum bilirubin, International Normalized Ratio (INR) >1.5 or prothrombin time (PT) >18 seconds
12. Any active local or systemic infection
13. Known heparin-induced thrombocytopenia
14. Known active bleeding disorder and/or any coagulopathy or thromboembolic disease
15. Allergies to study device (nitinol) or agents/medication, such as contrast agents or aspirin, that can't be controlled medically
16. Previous enrolment in this study
17. Subject is participating in another study
18. Pregnant or breastfeeding woman or woman in fertile period not taking adequate contraceptives
19. Any other condition which, in the judgement of the investigator would preclude adequate evaluation for the safety and performance of the study conduit

Intra-operative exclusion criteria:

1. Unsuitable anatomy to implant the XPAD conduit (e.g. target vessel diameter smaller than anticipated; severe calcification)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate | 12 months
  Primary patency: Defined as the interval between graft implantation and the first intervention to maintain or restore patency
Freedom from device-related SAE | Day 1, 1, 6 and 12 months

SECONDARY OUTCOMES:
Implantation success rate | Day 1
  Implantation success: Defined as a technically successful XPAD conduit implantation in the planned configuration, free from kinking and tension in the anastomoses, and a patent XPAD conduit at the moment of discharge
Freedom from Major Bleeding events | Day 1, 1 and 6 months
  Major Bleeding: Defined as type 3, 4 or 5 bleeding according to the Bleeding Academic Research Consortium (BARC) classifications
Patency (primary, primary assisted, and secondary) rates | 6, 12, 24, and 36 months
  Primary patency: Defined as the interval between graft implantation and the first intervention to maintain or restore patency.
  Assisted primary patency: Defined as the interval between graft implantation and the first occlusion (thrombosis), including interventions (operative or endovascular) aimed to maintain the functionality the graft.
  Secondary patency: Defined as the interval between graft implantation and abandonment with or without interventions (operative or endovascular) aimed to maintain the functionality the graft, including occurrence of a censored event (death, change of modality, loss of follow-up)
Freedom from device-related SAE | 24 and 36 months
Rate of wound/graft infections | 1, 6, 12, 24, and 36 months
Freedom from Major Amputations | 1, 6, 12, 24, and 36 months
  Major Amputation: Defined as any amputation that results in limb shortening
Freedom from all-cause mortality | 1, 6, 12, 24, and 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Investigación y Manejo del Cáncer (CIMCA), San José, Costa Rica